CLINICAL TRIAL: NCT03438045
Title: Implementing a Participatory, Multi-level Intervention to Improve Asian American Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU College of Dentistry (Other)
Collaborators: NYU School of Medicine (Unknown); State University of New York at Buffalo (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Mary E. Northridge, Associate Professor, NYU College of Dentistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: s17-01077; 1U56DE027447-01 (NIH)
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Results first posted 2021-07-06 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Oral Disease; Dental Caries
Keywords: Chinese American; implementation science; feasibility; acceptability; oral health; dental care; health equity; urban health
MeSH Terms: conditions — Mouth Diseases; Dental Caries

STUDY DESIGN:
Intervention Model Description: Feasibility and acceptability study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partnered Intervention (Experimental): The aspects of the partnering package of evidence-based intervention strategies are: (1) written agreements of collaboration for dental screening, health promotion, and incentives; (2) culturally-tailored and language-specific adaptation of materials; (3) demonstrations with role-playing of proper brushing with fluoride toothpaste and flossing techniques; and (4) CHW follow-up with patients of oral health care receipt and dental hygiene behaviors. Additionally, bilingual (English and Mandarin Chinese) CHWs will receive additional training in oral health promotion demonstration, oral health services and programs available at local clinics and hospitals, information about dental and health insurance, and evidence-based oral health behaviors.
  Interventions: Behavioral: Partnered intervention

INTERVENTIONS:
Behavioral: Partnered intervention — CHWs will provide dental education and counseling, lead interactive demonstrations of brushing with fluoride toothpaste and flossing, and improve access to dental care through dental coverage enrollment and linkage to local dentists.

SUMMARY:
This feasibility and acceptability study will be conducted at 3 community outreach centers serving an urban, low-income Chinese population. The study will evaluate the feasibility and acceptability of implementing a partnered intervention to improve the oral and general health of low-income, urban Chinese American adults and of using remote data entry into an electronic health record (EHR). The research staff will survey a sample of Chinese American patients screened at each center about their satisfaction with the partnered intervention and about their oral health behaviors. An additional sample selected from providers [dentists and community health workers (CHW)], research staff, New York University (NYU) administrators, site directors, and community advisory board (CAB) members will participate in structured interviews about the partnered intervention. The remote EHR evaluation will include group adaptation sessions and workflow analyses via multiple recorded sessions with research staff, NYU administrators, outreach site directors, and providers (dentists and CHWs). The study will also model knowledge held by these non-patient participants (including CAB members) to evaluate and enhance the partnered intervention during and/or after the feasibility and acceptability study for use in future implementations.

DETAILED DESCRIPTION:
Introduction: While the US health care system has the capability to provide amazing treatment of a wide array of conditions, this care is not uniformly available to all population groups. Oral health care is one of the dimensions of the US health care delivery system in which striking disparities exist. More than half of the population does not visit a dentist each year. Improving access to oral health care is a critical and necessary first step to improving oral health outcomes and reducing disparities. Fluoride has contributed profoundly to the improved dental health of populations worldwide and is needed regularly throughout the life course to protect teeth against dental caries. To ensure additional gains in oral health, fluoride toothpaste should be used routinely at all ages. Evidence-based guidelines for annual dental visits and brushing teeth with fluoride toothpaste form the basis of this implementation science project that is intended to bridge the care gap for underserved Asian American populations by improving access to quality oral health care and enhancing effective oral health promotion strategies. The ultimate goal of this study is to provide information for the design and implementation of a randomized controlled trial of a participatory, multi-level, partnered (i.e., with community stakeholders) intervention to improve the oral and general health of low-income Chinese American adults.

Methods: This study will evaluate the feasibility and acceptability of implementing a partnered intervention using remote data entry into an electronic health record (EHR) to improve access to oral health care and promote oral health. The research staff will survey a sample of Chinese American patients (planned n = 90) screened at 3 outreach centers about their satisfaction with the partnered intervention. Providers (dentists and community health workers), research staff, administrators, site directors, and community advisory board members will participate in structured interviews about the partnered intervention. The remote EHR evaluation will include group adaptation sessions and workflow analyses via multiple recorded sessions with research staff, administrators, outreach site directors, and providers. The study will also model knowledge held by non-patient participants to evaluate and enhance the partnered intervention for use in future implementations.

ELIGIBILITY:
Inclusion Criteria:

Outreach center patients will be enrolled into either or both of 2 groups.

Approximately 50 patients from each of 3 centers (n = 150) will be consented to allow their data to be entered via the remote EHR. These EHR patient participants must meet all of the following criteria to be enrolled:

1. Greater than or equal to 21 years of age
2. Self-identify as being of Chinese ethnicity
3. Live in any of the 5 boroughs of New York, NY and visit a participating outreach center
4. Able and willing to provide informed consent to have their data entered into the remote EHR

Approximately 30 patients from each of 3 centers (n = 90) will be consented to participate in an exit interview and a follow-up interviews. These interview patient participants must meet all of the following criteria:

1. Greater than or equal to 21 years of age
2. Self-identify as being of Chinese ethnicity
3. Live in any of the 5 boroughs of New York, NY and visit a participating outreach center
4. Able and willing to provide informed consent and participate in an exit interview and a follow-up interview

Approximately 20 research staff, NYU administrators, outreach center directors, and providers (dentists and CHWs) will be enrolled to participate in interviews about the partnered intervention and/or remote EHR. These non-patient participants must meet all of the following criteria:

1. Greater than or equal to 18 years of age
2. Be employed or volunteers at participating outreach centers or employed at NYU
3. For CHW-staff, speak and read Mandarin Chinese
4. Able and willing to provide informed consent

Approximately 32 non-patient participants (research staff, NYU administrators, CAB members, outreach site directors, and providers (dentists and CHWs) will be enrolled to participate in interviews and a group model-building workshop to inform model development by sharing their knowledge about factors that influence access to oral health care and care-seeking behaviors among low-income, urban Chinese American adults. These individuals must meet all of the following criteria:

1. Greater than 18 years of age
2. Be employed or volunteers at participating outreach centers or employed at NYU
3. Able and willing to provide informed consent

Exclusion Criteria:

Individuals meeting any of the following criteria will not be enrolled as either EHR patient participants or interview patient participants:

1. Have an acute or terminal illness or a serious mental illness or any other severe health condition(s) that might preclude visiting an oral health care provider
2. Are currently participating in another oral health study

Individuals meeting any of the following criteria will not be enrolled to complete the interviews about the partnered intervention or remote EHR or to provide input to the knowledge modeling activities:

1. Staff in functional areas that do not directly service patients (e.g., custodial staff) A patient participant may participate in either the EHR patient participant group only or both patient participant groups (interview patient participants are a subset of EHR patient participants). A non-patient participant may participate in any or all of the non-patient participant data collection activities. Co-participation in activities by any subject is not required.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa W Riddle, PhD, Study Chair — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- NYU College of Dentistry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Northridge ME, Metcalf SS, Yi S, Zhang Q, Gu X, Trinh-Shevrin C. A Protocol for a Feasibility and Acceptability Study of a Participatory, Multi-Level, Dynamic Intervention in Urban Outreach Centers to Improve the Oral Health of Low-Income Chinese Americans. Front Public Health. 2018 Feb 14;6:29. doi: 10.3389/fpubh.2018.00029. eCollection 2018. PMID 29492400
- [Result] Northridge ME, Kavathe R, Zanowiak J, Wyatt L, Singh H, Islam N. Implementation and dissemination of the Sikh American Families Oral Health Promotion Program. Transl Behav Med. 2017 Sep;7(3):435-443. doi: 10.1007/s13142-017-0466-4. PMID 28144833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five Chinese American community-based organizations have already volunteered to participate in this study:
  * Asian Americans for Equality.
  * Chinatown YMCA, a Branch of the YMCA of Greater New York.
  * Chinese American Planning Council.
  * Coalition for Asian American Children and Families.
  * Hamilton-Madison House.
  The three outreach centers for this study will be selected from among the affiliated outreach centers of these organizations.
Pre-assignment Details: No assignment to groups was part of this feasibility and acceptability study. All participants received the intervention.
Period: Overall Study
Arm/Group | Partnered Intervention
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The proposed study will enroll Chinese American adults aged 21 years and older.
Arm/Group | Partnered Intervention
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participants in years Population: Missing information for 1 participant.
  years
    number analyzed (Participants) | 74
    (all) | 58.9 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants] — We estimate that approximately 60% of our enrolled patient participants will be women, based on our experience with conducting community-based screening events. Population: Missing information for 1 participant.
  Participants
    number analyzed (Participants) | 74
    Female | 62
    Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The study population is Chinese American adults living in any of the five boroughs of New York, NY.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 74
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-identify as being of Chinese ethnicity (Asian race).
  Participants
    American Indian or Alaska Native | 0
    Asian | 74
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 75
Preferred language [Count of Participants; unit: Participants] — Chinese language (e.g., Mandarin, Cantonese)
  Participants
    Chinese | 74
    English | 0
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Agree or Strongly Agree With the Statement, "The Community Health Worker (CHW) Helped me to Improve How I Take Care of my Health" Based on a 4-point Likert Scale.
Description: Number of patients who agree or strongly agree with the statement that the CHW helped me to improve how I take care of my health, based on exit interviews administered via in-person paper questionnaire at the end of the outreach event (4 possible responses: strongly agree, agree, disagree, strongly disagree) used in the Sikh American Families Oral Health Promotion Program.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Partnered Intervention
Number analyzed (Participants) | 72
Participants
  Strongly agree | 21
  Agree | 50
  Disagree | 1
  Strongly disagree | 0

2. Secondary Outcome: Number of Patients Who Agree or Strongly Agree With the Statement, "The Community Health Worker (CHW) Answered my Questions or Concerns" Based on a 4-point Likert Scale.
Description: Number of patients who agree or strongly agree with the statement that the CHW answered my questions or concerns, based on exit interviews administered via in-person paper questionnaire at the end of the outreach event (4 possible responses: strongly agree, agree, disagree, strongly disagree) used in the Sikh American Families Oral Health Promotion Program.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Partnered Intervention
Number analyzed (Participants) | 67
Participants
  Strongly agree | 16
  Agree | 50
  Disagree | 1
  Strongly disagree | 0

3. Secondary Outcome: Number of Patients Who Agree or Strongly Agree With the Statement, "The Information and Topics Were Informative" Based on a 4-point Likert Scale.
Description: Number of patients who agree or strongly agree with the statement that the information and topics were informative, based on exit interviews administered via in-person paper questionnaire at the end of the outreach event (4 possible responses: strongly agree, agree, disagree, strongly disagree) used in the Sikh American Families Oral Health Promotion Program.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Partnered Intervention
Number analyzed (Participants) | 69
Participants
  Strongly agree | 17
  Agree | 52
  Disagree | 0
  Strongly disagree | 0

4. Secondary Outcome: Number of Patients Who Agree or Strongly Agree With the Statement, "The In-person Demonstrations Were Helpful in Improving Oral Health" Based on a 4-point Likert Scale.
Description: Number of patients who agree or strongly agree with the statement that the in-person demonstrations were helpful in improving oral health, based on exit interviews administered via in-person paper questionnaire at the end of the outreach event (4 possible responses: strongly agree, agree, disagree, strongly disagree) used in the Sikh American Families Oral Health Promotion Program.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Partnered Intervention
Number analyzed (Participants) | 69
Participants
  Strongly agree | 17
  Agree | 52
  Disagree | 0
  Stronly disagree | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: UPs that are serious adverse events will be reported to the IRB and to NIDCR within 1 week of the investigator becoming aware of the event.
Arm/Group | Partnered Intervention
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

LIMITATIONS AND CAVEATS:
A limitation of this pilot study is the small sample size, especially for completion of the 1-month follow-up phone calls. As of March 2020, all research activities were halted at New York University (NYU) in New York, NY, USA, so we ended enrollment on the current pilot study and analyzed the data at hand. Additional limitations of this research include potential recall bias regarding the retrospective assessments, and possible response bias associated with self-reported behaviors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03438045/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03438045/ICF_001.pdf